CLINICAL TRIAL: NCT06672250
Title: The Correlation Between Circulatory Tumor Cells and Venous Thrombosis
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsin-Fu Lee, Professor Attending Physicians, Chang Gung Memorial Hospital
Other Study IDs: 202400562B0
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Tumor Cells, Circulating; Venous Thrombosis
Keywords: Cancer; Thrombosis; Venous thromboembolism; Circulating tumor cells; Endovascular therapy
MeSH Terms: conditions — Neoplastic Cells, Circulating; Venous Thrombosis; Neoplasms; Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer for CTC culture: a thrombosis patient with cancer .
  Interventions: Procedure: CTCs/CTMs culture
- health for CTC culture: a thrombosis patient without cancer
  Interventions: Procedure: CTCs/CTMs culture

INTERVENTIONS:
Procedure: CTCs/CTMs culture — Collect the thrombosis from participants underwent catheter-based thrombectomy.To characterized by cancer-specific surface markers successfully and identify within the culture

SUMMARY:
Research indicates a strong correlation between cancer and thrombosis, with approximately 20% of blood clots in the U.S. being cancer-related, according to CDC data. Cancer patients face a 4-7 times higher risk of thrombosis compared to non-cancer individuals. Certain cancer treatments, such as chemotherapy and targeted therapy, elevate the likelihood of venous thromboembolism (VTE). Cancer patients with VTE exhibit a significantly higher hazard ratio (H.R.) of 3.4 compared to those without VTE.

This study aims to explore three main topics: (1) Comparing the differences and similarities of leukocyte populations between cancer-associated thrombosis (CAT) and venous thromboembolism (VTE). (2) Characterizing the factors contributing to increased incidence of cancer-associated thrombosis (CAT), with the hypothesis that circulating tumor microemboli (CTM) may express more thrombosis-related proteins than CTCs. (3) Understanding the effects of aspirin or NOACs on cancer-associated thrombosis and CTM formation.

DETAILED DESCRIPTION:
Research indicates a strong correlation between cancer and thrombosis, with approximately 20% of blood clots in the U.S. being cancer-related, according to CDC data. Cancer patients face a 4-7 times higher risk of thrombosis compared to non-cancer individuals. Certain cancer treatments, such as chemotherapy and targeted therapy, elevate the likelihood of venous thromboembolism (VTE). Cancer patients with VTE exhibit a significantly higher hazard ratio (H.R.) of 3.4 compared to those without VTE.

The mechanisms underlying cancer-related thrombosis are intricate. Cancer cells can directly activate coagulation and platelets through various factors, including tissue factor (T.F.), particularly prevalent in specific cancers like pancreatic and ovarian, correlating with a heightened VTE risk and poorer prognosis. Additionally, factors such as podoplanin (PDPN), plasminogen activation inhibitor-1 (PAI-1), and cancer procoagulant (C.P.) further promote coagulation. Inflammatory cytokines originating from tumor cells and cancer-derived factors stimulate neutrophil extracellular traps, contributing to thrombosis.

Metastatic tumors facilitate cancer cell dissemination and entry into blood vessels, leading to thrombosis in certain instances. Analyzing circulating tumor cells (CTCs) from biopsies aids in comprehending cancer metastasis and identifying treatment targets. However, isolating these rare CTCs from blood presents a challenge. Endovascular therapy has made strides in thrombosis treatment, with endovascular thrombectomy showing promise in severe thrombosis cases. It is proposed that aspirating thrombi during this procedure could yield CTCs for further examination regarding the impact of cancer cells on thrombogenesis.

This study aims to explore three main topics: (1) Comparing the differences and similarities of leukocyte populations between cancer-associated thrombosis (CAT) and venous thromboembolism (VTE). (2) Characterizing the factors contributing to increased incidence of cancer-associated thrombosis (CAT), with the hypothesis that circulating tumor microemboli (CTM) may express more thrombosis-related proteins than CTCs. (3) Understanding the effects of aspirin or NOACs on cancer-associated thrombosis and CTM formation.

ELIGIBILITY:
Inclusion Criteria:

1. age≧18
2. participants (1)participants without cancer: without cancer in five years (2)participants with cancer:pathology reveal have malignant tumor
3. patients who underwent catheter-based thrombectomy
4. agree do the thrombectomy

Exclusion Criteria:

1. participants without cancer (1).shock (2).severe sepsis (3).with cancer in five years
2. participants with cancer (1).shock (2).severe sepsis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who underwent catheter-based thrombectomy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
cell culture | baseline
  cancer-specific surface markers
RNA-seq | baseline
  DNA/RNA extraction of sorted cells as instruments' maneuvers and do the RNA-seq

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Fu Lee, PhD, Study Director — New Taipei City TuCheng Hospital
Locations (1):
- New Taipei City TuCheng Hospital, New Taipei City, Taiwan

REFERENCES:
- [Result] Falanga A, Russo L. Epidemiology, risk and outcomes of venous thromboembolism in cancer. Hamostaseologie. 2012;32(2):115-25. doi: 10.5482/ha-1170. Epub 2011 Oct 5. PMID 21971578